CLINICAL TRIAL: NCT05843227
Title: Description of the Organizational Measures Framing Surgery for Idiopathic Scoliosis in Children and Adolescents - Practice Survey
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN1322022/CHUSTE
Record Dates: First submitted 2023-03-14; First posted 2023-05-06 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Practice Scope
Keywords: pediatric orthopaedic surgeon; Idiopathic Scoliosis; Pediatric; Enhanced Rehabilitation After Surgery (ERAS); posterior vertebral arthrodesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- paediatric orthopaedic surgeons: paediatric orthopaedic surgeons in the national territory who routinely treat idiopathic scoliosis in children and adolescents and who are members of the Société Française d'Orthopédie Pédiatrique (SoFOP) will be included.
  questionnaire will be completed. .
  Interventions: Other: questionnaire on the organizational management

INTERVENTIONS:
Other: questionnaire on the organizational management — Data are collected through a questionnaire on the organizational management of the pre-operative / intraoperative / postoperative periods.

SUMMARY:
The pediatric orthopaedic surgeon treats idiopathic scoliosis in children and adolescents using the posterior vertebral arthrodesis technique. This surgery is considered "heavy" by the child and families while it is intended for a healthy population. Through this study to take stock of the measures governing idiopathic scoliosis surgery (pre-operative, intra-operative and post-operative) within the various pediatric orthopedic surgery departments on the French national territory.

DETAILED DESCRIPTION:
The goal is to measure the interest of harmonizing the preparation of orthopedic surgery for idiopathic scoliosis in children and adolescents by implementing a ERAS (Enhanced Rehabilitation After Surgery) protocol nationwide.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric orthopaedic surgeons in the national territory who routinely treat idiopathic scoliosis in children and adolescents and who are members of the Société Française d'Orthopédie Pédiatrique (SoFOP)

Exclusion Criteria:

* Refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Paediatric orthopaedic surgeons in the national territory who routinely treat idiopathic scoliosis in children and adolescents and who are members of the Société Française d'Orthopédie Pédiatrique (SoFOP) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-02-25 (Actual)

PRIMARY OUTCOMES:
practices currently in force for the preparation of posterior vertebral arthrodesis | Month: 3
  Analysis practices currently in force for the preparation of posterior vertebral arthrodesis by intern results questionnaires.
  questionnaire is created by the department specifically for this study

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Gautheron, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No